CLINICAL TRIAL: NCT02639455
Title: Survey of the Collective 16s rRNA Genes From Bacterial Populations From Exercising and Non-exercising Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2015-1268
Record Dates: First submitted 2015-12-01; First posted 2015-12-24 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Athlete group (No Intervention): Participants wo regularly exercise and are student athletes.
- Non-exercise group (No Intervention): Participants who are not student athletes.
- Exercise group (Experimental): Participants are not student athletes but commit to modest exercise for 5 weeks as part of this study.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Participants will exercise 4 days per week, 20 minutes per session for 5 weeks (a total of 400 minutes). Exercise will be independent (with the goal of 85% of max effort for at least 2 minutes each session) and consist of running, jumping jacks, sit ups, push ups, or burpees depending on the participant's comfort and skill.
  Arms: Exercise group

SUMMARY:
Poor oral health can greatly impact quality of life and can also impact overall health. For instance, research suggests that poor oral health may be associated with systemic diseases such as diabetes, heart disease, and stroke. Therefore, there is a need to investigate the causes of poor oral health.

The idea that athletes may have a propensity for dental caries has been gaining traction. There have been recent reports of high levels of dental caries, dental erosion and periodontal diseases among elite soccer players compared to the general public and in athletes from a wide range of sports. However, to date, no studies have investigated the oral microbiome of athletes.

Many factors affect the development of dental caries, including host factors, diet, and the microorganisms present in the oral cavity. More than 700 types of bacterial species have been detected in the oral cavity, and some have been identified to play a significant role in the development of oral disease. Streptococcus mutans is the main species involved in dental decay with various lactobacilli also involved in the disease process. Treponema denticola, Porphyromonas ginigivalis, and Aggregatibacter actinomycetemcomitans are the main species involved in periodontal disease. It is not currently known if changes in the collective oral microbiome foster or impede the development of these pathogens.

Complex microbe-host interactions occur to allow for the progression of oral disease, with host nutrition and hygiene playing a significant role. Endurance athletes widely consume a variety of sport drinks, gels, and energy bars for supplementation of electrolytes and carbohydrates. The consumption of these foods leads to pH drops in the oral cavity and may contribute to tooth erosion and demineralization. Oral disease may also be exacerbated by the fluid and electrolyte deficit that impedes saliva flow during exercise. However, several studies have failed to demonstrate a clear link between sports drinks and an increased risk of dental caries among athletes.

Dental caries are caused by microorganisms in the oral cavity. These microbes may be affected by host factors or nutrition in the progression of oral disease. Due to the documented prevalence of dental caries in athletes and the lack of clear connection between sports drinks and dental caries, the investigators propose to investigate any correlation that may exist between exercise and the oral microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between the ages of 18-24 and must be willing and healthy enough to start a modest exercise program if they are chosen, at random, to do so.

Exclusion Criteria:

* Pregnant women, minors, and people over the age of 24 are excluded from the study.
* Anyone with a heart condition or other health condition that is not safely able to initiate a modest exercise program are excluded from the study.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Changes in DNA sequence of the 16S rRNA gene of each member of the bacterial population in the oral cavity of each participant. | Baseline and 5 weeks
  Changes in DNA sequence of the 16S rRNA genes will be assessed at 5 weeks after an exercise intervention and and compared to baseline populations.

IPD SHARING:
Plan to Share IPD: Undecided
De-identified participant data may be made available within 12 months after completion of the study if the study is published.